CLINICAL TRIAL: NCT05175664
Title: TRacking Alzheimer´s Disease: a Study of Disease trajeCtory and Development of Diagnostic and Disease Stage biomarKers in AD (TRACK-AD)
Brief Title: Novel Diagnostic and Disease Stage Biomarkers in AD
Acronym: TRACK-AD
Status: Completed | Type: Observational
Sponsor: Danish Dementia Research Centre (Network)
Responsible Party: Sponsor
Other Study IDs: H-21040317
Record Dates: First submitted 2021-12-01; First posted 2022-01-04 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Neuro-Degenerative Diseases; Vascular Dementia; Dementia With Lewy Bodies; Healthy Controls
Keywords: Biomarkers; Pupillometry; Actigraphy; Blood-based biomarkers
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia, Vascular; Lewy Body Disease | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood: A total of 12 mL of blood will be collected at the study visits. Afterwards, the blood will be centrifuged and the serum, plasma and the white blood cells will be extracted. These samples will be stored in the Danish Dementia Biobank prior to analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- MCI: Patients suffering from mild cognitive impairment (MCI) due to Alzheimer's disease.
  Interventions: Other: Long-term study
- AD: Patients diagnosed with mild to moderate Alzheimer's disease (AD)
  Interventions: Other: Long-term study; Other: Cross-sectional study
- NDD: Patients under investigation of a neurodegenerative disease (NDD)
  Interventions: Other: Short-term study
- DLB: Patients diagnosed with Dementia with Lewy Bodies (DLB)
  Interventions: Other: Cross-sectional study
- VaD: Patients with vascular dementia (VaD)
  Interventions: Other: Cross-sectional study
- FTD: Frontotemporal dementia (FTD)
  Interventions: Other: Cross-sectional study
- NPH: Normal pressure hydrocephalus (NPH)
  Interventions: Other: Cross-sectional study
- Healthy Controls: Healthy Controls without brain disease
  Interventions: Other: Cross-sectional study

INTERVENTIONS:
Other: Long-term study — No intervention. Investigations: cognitive tests, blood samples, pupillometry, actigraphy, and FDG-PET/MR brain scan.
  Groups: AD; MCI
Other: Short-term study — No intervention. Investigations: blood samples and pupillometry.
  Groups: NDD
Other: Cross-sectional study — No intervention. Investigations: cognitive tests, pupillometry and actigraphy.
  Groups: AD; DLB; FTD; Healthy Controls; NPH; VaD

SUMMARY:
This study will investigate the efficacy of novel biomarkers, namely blood-based biomarkers, pupillometry and actigraphy to track and predict progression of Alzheimer's disease (AD). Furthermore, the study will investigate the diagnostic value of pupillometry and actigraphy for AD.

DETAILED DESCRIPTION:
This study consist of three sub-studies.

In study 1, participants diagnosed with mild cognitive impairment due to AD or mild to moderate AD will be followed for up to 24 months with repeated blood samples, pupillometry, actigraphy, cognitive tests and a control brain scan.

In study 2, patients under investigation of a neurodegenerative disease who have a planned lumbar puncture in the Memory clinic will be invited to this study. Participants will undergo pupillometry and blood samples two times approximately one and four weeks after the lumbar puncture.

In study 3, participants with a dementia diagnosis will undergo pupillometry and actigraphy at a single visit.

ELIGIBILITY:
1. Longitudinal study:

   Inclusion criteria:
   * MCI due to AD, or mild or moderate AD dementia according to the National Institute on Aging and Alzheimer's Association (NIA-AA) diagnostic criteria
   * Caregiver willing to participate as an informant
   * MMSE >19 at inclusion
   * Brain FDG-PET/MRI or FDG/PET-CT
   * Able to cooperate to the investigations and give informed consent

   Exclusion criteria:
   * Other neurological or psychiatric illness that may affect neurofilament light (NfL) levels (severe neuropathy, multiple sclerosis (MS), stroke within the last 3 months, Wernicke encephalopathy)
   * Diagnosis of previous or current major psychiatric disorder (schizophrenia, bipolar disorder, psychosis) within last 2 years
   * Excessive alcohol intake or substance abuse within the last 2 years
   * Ophthalmological disorders that may affect pupillometry
   * Participating in drug trials or other intervention trials
2. Short-term study:

   Inclusion criteria:
   * Patients under investigation of a neurodegenerative disease
   * MMSE >19
   * Scheduled lumbar puncture/lumbar puncture performed within the last week prior to inclusion
   * Written consent form to the Danish Dementia Biobank
   * Able to cooperate to the investigations

   Exclusion criteria:
   * Other neurological or psychiatric illness that may affect NfL levels (severe neuropathy, MS, stroke within the last 3 months, Wernicke encephalopathy)
   * Excessive alcohol intake or substance abuse within the last 2 years
   * Ophthalmological disorders that may affect pupillometry
   * Participating in drug trials or other intervention trials
3. Cross-sectional study:

Inclusion criteria - Patients:

* A diagnosis of a dementia disorder
* Caregiver willing to participate as an informant
* MMSE >15 at inclusion
* Able to cooperate to the investigations
* Able to give informed consent

Exclusion criteria - Patients:

* Diagnosis of previous or current major psychiatric disorder (schizophrenia, bipolar disorder, psychosis) within last 2 years
* Excessive alcohol intake or substance abuse within the last 2 years
* Other known brain disorder
* Ophthalmological disorders that may affect pupillometry
* Participating in drug trials or other intervention trials

Inclusion criteria - Healthy Controls:

* Able to cooperate to the investigations
* Normal cognition
* Age 50-90 year

Exclusion criteria - Healthy Controls:

* Diagnosis of previous or current major psychiatric disorder (schizophrenia, bipolar disorder, psychosis) within last 2 years
* Excessive alcohol intake or substance abuse within the last 2 years
* Other known brain disorder
* Ophthalmological disorders that may affect pupillometry

Ages: 30 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the longitudinal study (1) the investigators will include 100 patients diagnosed with mild cognitive impairment due to Alzheimer's disease or diagnosed with mild to moderate Alzheimer's disease. In the short-term study (2) the investigators will include 40 patients who are under investigation of a neurodegenerative disease. In the cross-sectional study (3) the investigatorswill include 50 patients with Alzheimer's disease, 50 healthy controls without brain disease, and 100 patients with other forms of dementia (dementia with Lewy body, vascular dementia, normal pressure hydrocephalus, frontotemporal dementia).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in CDR | Two years
  Clinical Dementia Rating (CDR), a clinical tool for grading the relative severity of dementia with scores ranging from 0 (no impairment) to 3 (severe impairment).

SECONDARY OUTCOMES:
Changes in MMSE | Two years
  Mini Mental Status Examination (MMSE), used to test global cognitive function
Changes in MR brain scan | 12 months
  Magnetic Resonance Imaging (MR), used to asses changes in volumetric measurements
FDG-PET brain scan | 12 months
  Fluorodeoxyglucose (FDG)-Positron Emission Tomography (PET) of the brain, used to asses changes in brain metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Frederikke Kragh Clemmensen, MD, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Copenhagen, Denmark; Mathias Holsey Gramkow, MD, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Copenhagen, Denmark; Kristian Steen Frederiksen, MD, PhD, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Copenhagen, Denmark; Steen Gregers Hasselbalch, DMSc, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Copenhagen, Denmark; Anja Hviid Simonsen, MSc Pharm PhD, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Danish Dementia Research Centre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clemmensen FK, Gramkow MH, Simonsen AH, Ashton NJ, Huber H, Blennow K, Zetterberg H, Waldemar G, Hasselbalch SG, Frederiksen KS. Short-term variability of Alzheimer's disease plasma biomarkers in a mixed memory clinic cohort. Alzheimers Res Ther. 2025 Jan 21;17(1):26. doi: 10.1186/s13195-024-01658-7. PMID 39838483